CLINICAL TRIAL: NCT02722980
Title: A Randomized, Double-blind, Placebo-controlled, Parallel-group Clinical Study Aiming to Evaluate the Efficacy on BMD and Safety of a Probiotic Product in a Population of Healthy Women in Early Post-menopausal Phase, During an Intervention Period of 12 Months
Brief Title: Efficacy of a Probiotic Product on Bone Mineral Density (BMD) in Healthy Women in Early Post-menopausal Phase
Acronym: ProBone16
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Probi AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: ProBone16
Record Dates: First submitted 2016-03-16; First posted 2016-03-30 (Estimated); Last update posted 2018-04-17 (Actual); Status verified 2018-04

CONDITIONS: Osteopenia
MeSH Terms: conditions — Bone Diseases, Metabolic | interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Capsules
  Interventions: Dietary Supplement: Placebo
- Active (Active Comparator): Capsules.
  Interventions: Dietary Supplement: : Probiotic capsules

INTERVENTIONS:
Dietary Supplement: Placebo — The intervention consists of capsules containing placebo.
  Arms: Placebo
Dietary Supplement: : Probiotic capsules — The intervention consists of capsules containing probiotics.
  Arms: Active

SUMMARY:
The aim of the current study is to evaluate the efficacy of a probiotic product on bone mineral density (BMD) in healthy early post-menopausal women, compared to placebo. The primary endpoint is to assess changes of BMD at lumbar spine after an intervention period of 12 months. Changes in BMD at the femoral neck (hip) will also be measured as well as changes in bone turnover markers during the period of 12 months.

ELIGIBILITY:
Inclusion Criteria:

For inclusion in the study, subjects must fulfil the following criteria:

1. Willing and able to give written informed consent for participation in the study.
2. Healthy women in early post-menopausal phase (at least two [2] years but a maximum of 12 years since the last menstruation and at least one [1] year since the last intake of hormone replacement therapy).
3. BMI ≥ 18 and ≤ 30 at screening.
4. BMD T-score in the lumbar spine (L1-L4) > -2.5, as measured by DXA.
5. Commitment not to use any products that may influence the study outcome in the opinion of the Investigator.
6. Ability to understand and comply with the requirements of the study, as judged by the Investigator.

Exclusion Criteria:

Subjects must not enter the study if any of the following exclusion criteria are fulfilled:

1. Relevant history of >1 previous fracture after 50 years of age, as judged by the Investigator.
2. T-score ≤ - 2.5, in the total hip or lumbar spine (L1-L4). These subjects should be forwarded to a GP for further investigation.
3. History of metabolic bone disease.
4. Unstable weight (± five [5] kg) during the last six (6) months.
5. History of hyperthyroidism or unstable hypothyroidism.
6. Diagnosed with disease causing secondary osteoporosis within the last year, including primary hyperparathyroidism, chronic obstructive pulmonary disease, inflammatory bowel disease (IBD), celiac disease or diabetes.
7. Known history of rheumatoid arthritis, clinically significant kidney or heart disease, as judged by the Investigator.
8. Gastric bypass surgery performed.
9. History of immunodeficiency or immunosuppressive treatment.
10. Chronic or acute diarrheal disease.
11. Recently diagnosed malignancy (within the last five [5] years).
12. Use of products containing probiotic bacteria (more than once per week) within four (4) weeks prior to baseline.
13. Per-oral use of corticosteroids.
14. Use of calcium and/or vitamin D supplements within one (1) month prior to baseline.
15. Use of any anti-resorptive therapy, including e.g. systemic hormone replacement therapy, bisphosphonates (currently or during last 12 months)
16. Use of any bone-formation stimulating therapy (currently or during the last 12 months).
17. Use of antibiotics during the last two (2) months.
18. Frequent user of antibiotics (>2 courses during the last 12 months) due to inter-current infection episodes.
19. Smoking or use of nicotine-containing products (currently or during the last six [6] months).
20. History of alcohol abuse, or excessive intake of alcohol, as judged by the Investigator.
21. Consumption of alcohol within 24 hours prior to the Baseline Visit.
22. Participation in any other clinical interventional study during the last three (3) months.
23. History of any clinically significant disease or disorder which, in the opinion of the Investigator, may either put the subject at risk because of participation in the study, or influence the results or the subject's ability to participate in the study
24. Known hypersensitivity to any of the ingredients in the IP or the placebo (maltodextrin, silicon dioxide, capsule [hypromellose, water] ± bacterial culture).
25. Blood or plasma donation within three (3) months prior to baseline.

Ages: 45 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 249 (Actual)
Dates: Start 2016-04; Primary Completion 2018-01 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Change in BMD at lumbar spine following an intervention period of 12 months and measured by DXA. | Change in BMD from baseline to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Dan Curiac, Principal Investigator — Gothenburg
Locations (2):
- Sweden (2):
  - Gothenburg
  - Uppsala

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jansson PA, Curiac D, Lazou Ahren I, Hansson F, Martinsson Niskanen T, Sjogren K, Ohlsson C. Probiotic treatment using a mix of three Lactobacillus strains for lumbar spine bone loss in postmenopausal women: a randomised, double-blind, placebo-controlled, multicentre trial. Lancet Rheumatol. 2019 Nov;1(3):e154-e162. doi: 10.1016/S2665-9913(19)30068-2. Epub 2019 Oct 23. PMID 38229392